CLINICAL TRIAL: NCT00751842
Title: A Phase III, 3-Arm, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Investigate the Impact of Diamyd on the Progression of Diabetes in Patients Newly Diagnosed With Type 1 Diabetes Mellitus (USA)
Brief Title: A Phase III Study to Investigate the Impact of Diamyd in Patients Newly Diagnosed With Type 1 Diabetes (USA)- DIAPREVENT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on other clinical trial results it was unlikely the study would meet the efficacy endpoints
Sponsor: Diamyd Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D/P3/07/5
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes; Juvenile Diabetes; Diabetes type 1; Autoimmune Diabetes; Insulin dependent Diabetes; Type 1 diabetes; Type 1 diabetes mellitus; Diamyd; rhGAD65; GAD; GAD-alum
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): This arm will receive 2 subcutaneous injections with 20 µg Diamyd on days 1 and 30, i.e., 1 prime and 1 booster dose, followed by 2 additional single doses with Diamyd 20 µg on days 90 and 270.
  Interventions: Drug: rhGAD65
- B (Active Comparator): This arm will receive 2 subcutaneous injections with 20 µg Diamyd on days 1 and 30, i.e., 1 prime and 1 booster dose, followed by 2 additional single doses with placebo on days 90 and 270.
  Interventions: Drug: rhGAD65
- C (Placebo Comparator): This arm will receive 4 injections of placebo, 1 each on days 1, 30, 90 and 270.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhGAD65 — Diamyd (rhGAD65) 20 µg injected subcutaneously at days 1, 30, 90 and 270.
  Arms: A
Drug: rhGAD65 — Diamyd (rhGAD65) 20 µg injected subcutaneously at days 1 and 30, followed by placebo injections at days 90 and 270.
  Arms: B
Drug: Placebo — Placebo injected subcutaneously at days 1, 30, 90 and 270.
  Arms: C

SUMMARY:
The intended purpose of this study was to determine whether Diamyd (rhGAD65 formulated in alum) is effective in preserving the body's own insulin producing capacity in patients recently diagnosed with type 1 diabetes.

Based on results from other clinical trials with the study drug it was judged unlikely this study would meet the intended primary or secondary efficacy endpoints. Therefore the primary focus of this study was changed to ensure that safety data was available for at least 6 months following the last dose of active study drug. Thereafter the study was terminated.

ELIGIBILITY:
Main Inclusion Criteria:

* Insulin dependent type 1 diabetes mellitus diagnosed within the previous 3 months at time of screening
* Fasting C-peptide level at time of screening above 0.1 nmol/L
* Elevated GAD65 antibodies (GADA) at time of screening
* Male and female patients between 10 and 20 years of age

Main Exclusion Criteria:

* Treatment with immunosuppressants or any anti-diabetic medications other than insulin
* A history of certain diseases or conditions (e.g. anemia, HIV, hepatitis, epilepsy, head trauma, neurological diseases or cerebrovascular accident, alcohol or drug abuse etc)
* Treatment with any vaccine within 1 month prior to planned first Diamyd dose or planned treatment with vaccine up to 2 months after the last injection with Diamyd, excluding the influenza vaccine
* Participation in other clinical trials with a new chemical entity within the previous 3 months
* Pregnancy or planned pregnancy within 1 year after the last Diamyd dose
* Presence of associated serious disease or condition which in the opinion of the investigator makes the patient non-eligible for the study

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 331 (Actual)
Dates: Start 2008-09; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Meal Stimulated C-peptide (area under the curve) | 15 months

SECONDARY OUTCOMES:
HbA1c | 15 months
Insulin Dose | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Palmer, Professor, Principal Investigator — University of Washington
Locations (43):
- United States (43):
  - University of Arizona, Tucson, Arizona
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Alex Endocrine Associates, Rogers, Arkansas
  - Children's Hospital Orange County, Orange, California
  - Rady Children's Hospital, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Christina Care Research institute, Newark, Delaware
  - University of Florida, Gainsville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital Research Institute, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - University of Iowa Hospitals and Clinicals, Iowa City, Iowa
  - Mid America Diabetes Associates, Wichita, Kansas
  - University of Kentucky College of Medicine, Lexington, Kentucky
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Children's Hospital, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Alzohaili Medical Consultants, Dearborn, Michigan
  - The Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Creighton Diabetes Center, Omaha, Nebraska
  - Kathryn Eckert, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Naomi Berrie Diabetes Center of Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Institute for Human Performance, Syracuse, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - University of Oklahoma, Schustermann Center Clinic, Tulsa, Oklahoma
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Regional Medical Clinic - Endocrinology, Rapid City, South Dakota
  - LeBonheur Children's Medical Center, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - CHRISTUS Santa Rosa Children's Hospital, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Benaroya Research Institute, Seattle, Washington

REFERENCES:
- [Background] Ludvigsson J, Faresjo M, Hjorth M, Axelsson S, Cheramy M, Pihl M, Vaarala O, Forsander G, Ivarsson S, Johansson C, Lindh A, Nilsson NO, Aman J, Ortqvist E, Zerhouni P, Casas R. GAD treatment and insulin secretion in recent-onset type 1 diabetes. N Engl J Med. 2008 Oct 30;359(18):1909-20. doi: 10.1056/NEJMoa0804328. Epub 2008 Oct 8. PMID 18843118
- [Background] Ludvigsson J, Krisky D, Casas R, Battelino T, Castano L, Greening J, Kordonouri O, Otonkoski T, Pozzilli P, Robert JJ, Veeze HJ, Palmer J, Samuelsson U, Elding Larsson H, Aman J, Kardell G, Neiderud Helsingborg J, Lundstrom G, Albinsson E, Carlsson A, Nordvall M, Fors H, Arvidsson CG, Edvardson S, Hanas R, Larsson K, Rathsman B, Forsgren H, Desaix H, Forsander G, Nilsson NO, Akesson CG, Keskinen P, Veijola R, Talvitie T, Raile K, Kapellen T, Burger W, Neu A, Engelsberger I, Heidtmann B, Bechtold S, Leslie D, Chiarelli F, Cicognani A, Chiumello G, Cerutti F, Zuccotti GV, Gomez Gila A, Rica I, Barrio R, Clemente M, Lopez Garcia MJ, Rodriguez M, Gonzalez I, Lopez JP, Oyarzabal M, Reeser HM, Nuboer R, Stouthart P, Bratina N, Bratanic N, de Kerdanet M, Weill J, Ser N, Barat P, Bertrand AM, Carel JC, Reynaud R, Coutant R, Baron S. GAD65 antigen therapy in recently diagnosed type 1 diabetes mellitus. N Engl J Med. 2012 Feb 2;366(5):433-42. doi: 10.1056/NEJMoa1107096. PMID 22296077
- [Background] Wherrett DK, Bundy B, Becker DJ, DiMeglio LA, Gitelman SE, Goland R, Gottlieb PA, Greenbaum CJ, Herold KC, Marks JB, Monzavi R, Moran A, Orban T, Palmer JP, Raskin P, Rodriguez H, Schatz D, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet GAD Study Group. Antigen-based therapy with glutamic acid decarboxylase (GAD) vaccine in patients with recent-onset type 1 diabetes: a randomised double-blind trial. Lancet. 2011 Jul 23;378(9788):319-27. doi: 10.1016/S0140-6736(11)60895-7. Epub 2011 Jun 27. PMID 21714999